CLINICAL TRIAL: NCT00103922
Title: A Randomized, 24-week, Double-blind, Placebo-controlled, Parallel-group Study to Evaluate the Efficacy, Safety and Tolerability of ARIFLO® (15mg BID) in Patients With Chronic Obstructive Pulmonary Disease (COPD)
Brief Title: Study In Subjects With COPD (Chronic Obstructive Pulmonary Disease)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CIL103657
Record Dates: First submitted 2005-02-17; First posted 2005-02-18 (Estimated); Last update posted 2016-10-28 (Estimated); Status verified 2016-10

CONDITIONS: Pulmonary Disease, Chronic Obstructive
Keywords: smokers cough
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Cilomilast

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm 1 (Experimental)
  Interventions: Drug: cilomilast

INTERVENTIONS:
Drug: cilomilast

SUMMARY:
This study was designed to determine if the investigational drug is effective and safe in individuals with COPD (chronic pulmonary disease)

ELIGIBILITY:
Inclusion criteria:

* Diagnosis of COPD and a history of cigarette smoking.

Exclusion criteria:

* Significant heart or lung disease not associated with COPD.
* Significant stomach or intestinal disease.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Actual)
Dates: Start 2004-11; Primary Completion 2007-01 (Actual); Study Completion 2007-01 (Actual)

PRIMARY OUTCOMES:
measure of lung function and quality of life in patients with COPD

SECONDARY OUTCOMES:
exacerbations in patients with COPD

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (106):
- United States (106):
  - GSK Investigational Site, Birmingham, Alabama
  - GSK Investigational Site, Jasper, Alabama
  - GSK Investigational Site, Phoenix, Arizona
  - GSK Investigational Site, Tempe, Arizona
  - GSK Investigational Site, Berkeley, California
  - GSK Investigational Site, Carmichael, California
  - GSK Investigational Site, Fullerton, California
  - GSK Investigational Site, Long Beach, California
  - GSK Investigational Site, Los Angeles, California
  - GSK Investigational Site, Murrieta, California
  - GSK Investigational Site, Rancho Mirage, California
  - GSK Investigational Site, Riverside, California
  - GSK Investigational Site, Sacramento, California
  - GSK Investigational Site, San Diego, California
  - GSK Investigational Site, San Jose, California
  - GSK Investigational Site, Sepulveda, California
  - GSK Investigational Site, Stockton, California
  - GSK Investigational Site, Torrance, California
  - GSK Investigational Site, Vista, California
  - GSK Investigational Site, Walnut Creek, California
  - GSK Investigational Site, Boulder, Colorado
  - GSK Investigational Site, Colorado Springs, Colorado
  - GSK Investigational Site, Denver, Colorado
  - GSK Investigational Site, Englewood, Colorado
  - GSK Investigational Site, Fort Collins, Colorado
  - GSK Investigational Site, Wheat Ridge, Colorado
  - GSK Investigational Site, Hartford, Connecticut
  - GSK Investigational Site, Stamford, Connecticut
  - GSK Investigational Site, Waterbury, Connecticut
  - GSK Investigational Site, Aventura, Florida
  - GSK Investigational Site, Brandon, Florida
  - GSK Investigational Site, DeLand, Florida
  - GSK Investigational Site, Fort Lauderdale, Florida
  - GSK Investigational Site, Largo, Florida
  - GSK Investigational Site, Longwood, Florida
  - GSK Investigational Site, Melbourne, Florida
  - GSK Investigational Site, Panama City, Florida
  - GSK Investigational Site, Pensacola, Florida
  - GSK Investigational Site, Tamarac, Florida
  - GSK Investigational Site, Tampa, Florida
  - GSK Investigational Site, West Palm Beach, Florida
  - GSK Investigational Site, Atlanta, Georgia
  - GSK Investigational Site, Decatur, Georgia
  - GSK Investigational Site, Coeur d'Alene, Idaho
  - GSK Investigational Site, Normal, Illinois
  - GSK Investigational Site, Evansville, Indiana
  - GSK Investigational Site, South Bend, Indiana
  - GSK Investigational Site, Wichita, Kansas
  - GSK Investigational Site, Madisonville, Kentucky
  - GSK Investigational Site, Lafayette, Louisiana
  - GSK Investigational Site, New Orleans, Louisiana
  - GSK Investigational Site, Slidell, Louisiana
  - GSK Investigational Site, Sunset, Louisiana
  - GSK Investigational Site, Boston, Massachusetts
  - GSK Investigational Site, Cadillac, Michigan
  - GSK Investigational Site, Minneapolis, Minnesota
  - GSK Investigational Site, Jefferson City, Missouri
  - GSK Investigational Site, Saint Charles, Missouri
  - GSK Investigational Site, St Louis, Missouri
  - GSK Investigational Site, Billings, Montana
  - GSK Investigational Site, Missoula, Montana
  - GSK Investigational Site, Las Vegas, Nevada
  - GSK Investigational Site, Cherry Hill, New Jersey
  - GSK Investigational Site, Bronxville, New York
  - GSK Investigational Site, Cortland, New York
  - GSK Investigational Site, Larchmont, New York
  - GSK Investigational Site, New York, New York
  - GSK Investigational Site, Chapel Hill, North Carolina
  - GSK Investigational Site, Charlotte, North Carolina
  - GSK Investigational Site, Elizabeth City, North Carolina
  - GSK Investigational Site, High Point, North Carolina
  - GSK Investigational Site, Statesville, North Carolina
  - GSK Investigational Site, Chardon, Ohio
  - GSK Investigational Site, Columbus, Ohio
  - GSK Investigational Site, Dayton, Ohio
  - GSK Investigational Site, Sylvania, Ohio
  - GSK Investigational Site, Lake Oswego, Oregon
  - GSK Investigational Site, Medford, Oregon
  - GSK Investigational Site, Portland, Oregon
  - GSK Investigational Site, Allentown, Pennsylvania
  - GSK Investigational Site, Downington, Pennsylvania
  - GSK Investigational Site, Elverson, Pennsylvania
  - GSK Investigational Site, Erie, Pennsylvania
  - GSK Investigational Site, Pittsburgh, Pennsylvania
  - GSK Investigational Site, Swarthmore, Pennsylvania
  - GSK Investigational Site, East Providence, Rhode Island
  - GSK Investigational Site, Charleston, South Carolina
  - GSK Investigational Site, Gaffney, South Carolina
  - GSK Investigational Site, Greer, South Carolina
  - GSK Investigational Site, Simpsonville, South Carolina
  - GSK Investigational Site, Spartanburg, South Carolina
  - GSK Investigational Site, Bristol, Tennessee
  - GSK Investigational Site, Chattanooga, Tennessee
  - GSK Investigational Site, Johnson City, Tennessee
  - GSK Investigational Site, Knoxville, Tennessee
  - GSK Investigational Site, Corsicana, Texas
  - GSK Investigational Site, Dallas, Texas
  - GSK Investigational Site, Fort Worth, Texas
  - GSK Investigational Site, San Antonio, Texas
  - GSK Investigational Site, Salt Lake City, Utah
  - GSK Investigational Site, Richmond, Virginia
  - GSK Investigational Site, Bellingham, Washington
  - GSK Investigational Site, Spokane, Washington
  - GSK Investigational Site, Tacoma, Washington
  - GSK Investigational Site, Morgantown, West Virginia
  - GSK Investigational Site, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Statistical Analysis Plan: CIL103657 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: CIL103657 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: CIL103657 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: CIL103657 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: CIL103657 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: CIL103657 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register